CLINICAL TRIAL: NCT02312349
Title: Assessment of Gluten-Free Availability in Elaborated Food Stores in Three Neighbourhoods of Buenos Aires City
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Universidad Isalud (Unknown)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1770
Record Dates: First submitted 2014-12-03; First posted 2014-12-09 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Gluten free elaborated food
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Celiac disease (CD) is a chronic autoimmune disorder in genetically susceptible individuals characterized by inflammation of the small intestine due to gluten intolerance. This protein is found in cereals such as wheat, barley and rye. In Argentina, oats are also considered a toxic grain since are as highly contaminated as the previous three. For this reason, the acronym TACC (Trigo, avena, cebada y centono: wheat, oats, barley and centono) is used for their identification. An effective treatment for celiac disease consists in a gluten-free diet (GFD). For most patients, a gluten-free intake results in a symptomatic and pathological complete remission and decreases the risk of complications.

The overall prevalence of CD is around 1% in several Western countries. An Argentinian study shows a 1.167 prevalence of CD in studied patients, being doubled for women than men. Another study in a closed population of the Health Plan of Hospital Italiano de Bs As estimated a prevalence of 0.22 CD diagnosis. In developed countries, for each diagnosed case there is an average of 5-10 cases that have not been diagnosed yet.

CD patients and their families should be properly informed about GFD, since there are many factors, voluntary and involuntary, which can affect the treatment. Even though a strict diet is imperative, food handling awareness is equally important in order to prevent cross-contamination and gluten intake hidden in certain products.

In recent years, several countries have shown an increasing interest in improving the supply of gluten-free foods in supermarkets, food factories and restaurants. In turn, a British study shows that chefs have less awareness about celiac disease than the overall population. Another Canadian study, which assessed the quality of life of people with CD, revealed that 80% of them avoid eating in restaurants for fear of contamination, causing a decrease in their social life.

In Argentina, there are associations that generate lists of marks and gluten-free products allowing safe intake of processed foods, however, it is unknown the food supply suitable for consumption for people with CD as well as the staff's knowledge in gluten-free food preparation in restaurants, pubs, pizzerias and fast food places. U.S. has quality assurance systems that certify good manufacturing practices and GFD handling in restaurants and selling local foods, although its application is not mandatory. In our country, there is no such certification, so food safety on restaurants can not be guaranteed.

Eating behaviors are influenced by the reality in which people live, including food availability indoors and outdoors. The current lifestyle leads more and more people to make meals away from home, so that the variety and quality of food sold in restaurants and other stores conditions the consumption. Thus, the availability of "safe" foods in places where people with CD carried some of their meals, help improve adherence to the GFD.

The aim of this study is to investigate gluten-free products' supply in elaborated food stores in Buenos Aires City and to discover the level of information possessed by manufacturers in the production of food.

ELIGIBILITY:
Inclusion Criteria:

- Restaurants, bars, pizzerias and fast food outlets, located in the three selected districts.

Exclusion Criteria:

-Refusal by the owner or manager of local participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It will generate a stratified random sample of 15% of businesses (restaurants, bars, pizzerias and fast food outlets) located in the three selected districts. To be used to sample a sampling frame of the selected districts conducted by the same research group (NCT01388972).
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Gluten Free elaborated food | At baseline
  Percentage of any available elaborated food free of gluten in its preparation an components for each restaurant evaluated

SECONDARY OUTCOMES:
Knowledge about Celiac Disease | At baseline
  Direct structure questionnaire about specific items related to knowledge about celiac disease directed to every person involved in storage, preparation or delivery of elaborated food
Appropriate preparation, delivery and storage of Gluten Free dishes | At baseline
  Direct evaluation by inspection of the complete process of storage, preparation or delivery of elaborated food in each restaurant to detect potential sources of gluten contamination

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Garipe LY, Bravo B, Fernandez M, Garcia M, Petrosini A, Soriano MM, Perman GP, Giunta DH. Evaluacion de la oferta de alimentos libres de gluten en locales de comida elaborada en la Ciudad Autonoma de Buenos Aires. Acta Gastroenterol Latinoam. 2015 Sep;45(3):190-7. Spanish. PMID 28590109